CLINICAL TRIAL: NCT00834288
Title: A Study to Compare the Bioavailability of Two Tramadol Hydrochloride Tablet Products (50 mg and 200 mg, Respectively) at Steady-state Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Labopharm Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MDT1-009
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2009-10-19 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Healthy Subjects; Pharmacokinetics; Bioavailability
Keywords: Healthy subjects; Pharmacokinetics; Bioavailability
MeSH Terms: interventions — Tramadol

ARMS (2):
- 1: 1x200 mg Tramadol HCl OAD tablet daily (Experimental)
  Interventions: Drug: Tramadol HCl
- 2: 1x50 mg Tramadol HCl IR (Ultram®) tablet 6-hourly (Active Comparator)
  Interventions: Drug: Tramadol HCl

INTERVENTIONS:
Drug: Tramadol HCl — 1x200 mg Tramadol HCl OAD tablet daily
  Arms: 1: 1x200 mg Tramadol HCl OAD tablet daily
Drug: Tramadol HCl — 1x50 mg Tramadol HCl IR (Ultram®) tablet 6-hourly
  Arms: 2: 1x50 mg Tramadol HCl IR (Ultram®) tablet 6-hourly

SUMMARY:
The purpose of this study was to compare the pharmacokinetic profiles at steady-state of the test product, Tramadol HCl Once-A-Day (OAD) 200 mg tablets and the reference product, Tramadol HCl 50 mg (IR) tablets (Ortho-McNeil Ultram®). For this purpose, the extent of absorption of tramadol and formation of O-desmethyltramadol (measures of systemic exposure) after multiple administration of 50 mg 6-hourly at 07:30, 13:30, 19:30 and 01:30 (reference product) and 200 mg 24-hourly at 07:30 (test product), were compared.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking, male and female subjects between the ages 18 to 55 years (inclusive).
* Body mass within 10% of the ideal mass in relation to height and age, according to the BMI
* Body mass not less than 70 kg.
* Findings within the range of clinical acceptability in medical history and physical examination, and laboratory results with the "normal ranges" for the relevant laboratory tests (unless the clinical investigator considers the deviation to be irrelevant for the purpose of the study).
* Normal ECG and vital signs, or abnormalities which the clinical investigator did not consider a disqualification for participation in the study
* Willingness to undergo a pre-study physical examination and pre- and post-study laboratory investigations.
* Ability to comprehend and willingness to sign both statements of Informed Consent (for screening and phase-related procedures)
* Non-smokers or past smokers who stopped smoking at least three months before entering the study
* For females, the following conditions had to be met:

  * had been postmenopausal for at least two years, or
  * had been surgically sterilized, or
  * was of childbearing potential, and all of the following conditions were met:
  * had a normal menstrual flow within one month before study entry, and
  * had negative urine pregnancy test at screening and on Day 1 of each study period. If the result of either test was positive, the subject would have been excluded from the study before receiving study medication.
  * had to agree to use an accepted method of contraception. The subject had to agree to continue with the same method throughout the study. Hormonal contraceptives were not allowed.

Exclusion Criteria:

* Evidence of psychiatric disorder, antagonistic personality, poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
* History of, or current compulsive alcohol abuse (> 10 drinks weekly), or regular exposure to other substances of abuse.
* Use of any medication, prescribed or over-the-counter, within 2 weeks prior to the first administration of study medication except if this would not have affected the outcome of the study in the opinion of the clinical investigator. Use of hormonal contraceptives agents by females was not allowed.
* Participation in another study with an experimental drug within 8 weeks before the first administration of study medication.
* Treatment within the previous 3 months with any drug with a well-defined potential for adversely affecting a major organ or system with evidence to this effect.
* Major illness during the 3 months before commencement of the screening period.
* History of hypersensitivity to the study drug or any related drugs.
* History of bronchial asthma.
* History of epilepsy.
* Relevant history or laboratory or clinical findings indicative of acute or chronic disease, likely to influence study outcome.
* Donation or loss of blood equal to or exceeding 500 ml during the 8 weeks before the first administration of study medication.
* Diagnosis of hypotension made during the screening period.
* Diagnosis of hypertension made during the screening period or current diagnosis of hypertension.
* Resting pulse of > 100 beats per minutes or < 45 beats per minutes during the screening period, either supine or standing.
* Positive testing for hepatitis B antigen.
* Significant liver disease, defined as active hepatitis or elevated liver enzymes (e.g., AST, ALT) > 3 times the upper boundary of the normal range.
* Positive urine screen for drugs of abuse.
* Positive urine screen for tobacco use.
* History of marijuana, barbiturates, amphetamine, or narcotic abuse within 12 months prior to study start.
* Previous participation in a tramadol study.
* pregnancy or lactation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2003-06; Primary Completion 2003-08 (Actual)

REFERENCES:
- [Result] Karhu D, Fradette C, Potgieter MA, Ferreira MM, Terblanche J. Comparative pharmacokinetics of a once-daily tramadol extended-release tablet and an immediate-release reference product following single-dose and multiple-dose administration. J Clin Pharmacol. 2010 May;50(5):544-53. doi: 10.1177/0091270009347673. Epub 2010 Jan 5. PMID 20051587
- See also: Approved labelling — http://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?id=9048

RESULTS

PARTICIPANT FLOW:
Groups:
- Test (Tramadol HCl OAD 200 mg) First: 1 x 200 mg Tramadol OAD (Once-A-Day) Tablet Daily test product dosed in first period followed by Tramadol IR (Ultram®) 50 mg 6-hourly) reference product dosed in the second period. The two treatment phases each started with a run-in period of 4 days (Days 1 to 4), a profile period and clinic stay of 3 days (Days 5 to 7) (clinic days and observation period) and a drug-free period of 16 days between treatment phases (Day 7 of Treatment phase I until Day 1 of the run-in period of Treatment phase II).
- Reference (Trazodone IR (Desyrel®) 100 mg 8-hourly) First: 1 x 100 mg Trazodone HCl IR (Desyrel®) Tablet 8-Hourly reference product dosed in first period followed by Trazodone OAD (Once-A-Day) Tablet Daily test product dosed in the second period. The two periods were separated by a washout of at least 7 calendar days.
  IR = Immediate Release.
Period: Treatment Phase I
Arm/Group | Test (Tramadol HCl OAD 200 mg) First | Reference (Trazodone IR (Desyrel®) 100 mg 8-hourly) First
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0
Period: Treatment Phase II
Arm/Group | Test (Tramadol HCl OAD 200 mg) First | Reference (Trazodone IR (Desyrel®) 100 mg 8-hourly) First
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Reference (Tramadol IR (Ultram®) 50 mg 6-hourly) First: 1 x 50 mg Tramadol HCl IR (Ultram®) Tablet 6-Hourly reference product dosed in first period followed by Tramadol OAD (Once-A-Day) Tablet Daily test product dosed in the second period. The two treatment phases each started with a run-in period of 4 days (Days 1 to 4), a profile period and clinic stay of 3 days (Days 5 to 7) (clinic days and observation period) and a drug-free period of 16 days between treatment phases (Day 7 of Treatment phase I until Day 1 of the run-in period of Treatment phase II). IR = Immediate Release.
- Total: Total of all reporting groups
Arm/Group | Test (Tramadol HCl OAD 200 mg) First | Reference (Tramadol IR (Ultram®) 50 mg 6-hourly) First | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 13 | 13 | 26.0
  >=65 years | 0 | 0 | 0.0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4.0
  Male | 11 | 11 | 22.0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Data Pairs at Steady State (AUCss)
Description: Area under the plasma concentration versus time data pairs over 24 hours (24h) at steady state, on day 5.
  ss = steady state. AUCss is also known as AUCtau.
Time Frame: 24 hours (day 5)
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Tramadol HCl OAD 200 mg: Tramadol HCl OAD 200 mg Group includes the treatment period 1 data from subjects in the "Test (Tramadol HCl OAD 200 mg) First" treatment sequence and the treatment period 2 data from subjects in the "Reference (Tramadol IR (Ultram®) 50 mg 6-hourly) First" treatment sequence.
- Tramadol IR (Ultram®) 50 mg 6-hourly: Tramadol IR (Ultram®) 50 mg 6-hourly Group includes the treatment period 1 data from subjects in the "Reference (Tramadol IR (Ultram®) 50 mg 6-hourly) First" treatment sequence and the treatment period 2 data from subjects in the "Test (Tramadol HCl OAD 200 mg) First" treatment sequence.
Arm/Group | Tramadol HCl OAD 200 mg | Tramadol IR (Ultram®) 50 mg 6-hourly
Number analyzed (Participants) | 26 | 26
ng*h/mL | 5991 (1330) | 6399 (1766)

2. Secondary Outcome: Maximum Plasma Concentration at Steady State(Cmax,ss)
Description: Maximum plasma concentration over 24 hours (24h) at steady state, on day 5. ss = steady state.
Time Frame: 24 hours (day 5)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tramadol HCl OAD 200 mg | Tramadol IR (Ultram®) 50 mg 6-hourly
Number analyzed (Participants) | 26 | 26
ng/mL | 345 (73) | 423 (97)

3. Secondary Outcome: Minimum Plasma Concentration at Steady State(Cmin,ss)
Description: Minimum plasma concentration over 24 hours (24h) at steady state on day 5. ss = steady state.
Time Frame: 24 hours (day 5)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tramadol HCl OAD 200 mg | Tramadol IR (Ultram®) 50 mg 6-hourly
Number analyzed (Participants) | 26 | 26
ng/mL | 157 (48) | 190 (64)

4. Secondary Outcome: Time to Peak Exposure (Tmax)
Description: Time to peak exposure over 24 hours (24h) at steady state on day 5.
Time Frame: 24 hours (day 5)
Measure: Median (Full Range); unit: hours
Arm/Group | Tramadol HCl OAD 200 mg | Tramadol IR (Ultram®) 50 mg 6-hourly
Number analyzed (Participants) | 26 | 26
hours | 4 [3 to 9] | 1 [1 to 3]

5. Secondary Outcome: Percentage Peak-trough Fluctuation (% PTF)
Description: Percentage peak-trough fluctuation over 24 hours (24h) at steady state on day 5.
  Percent peak-to-trough fluctuation is calculated as (Cmax - Cmin)/Cav*100, where Cmax is the maximum observed concentration, Cmin is the minimum observed concentration and Cav is the average concentration over 24 hours (where Cav = AUCss/24).
Time Frame: 24 hours (day 5)
Measure: Mean (Standard Deviation); unit: percentage of fluctuation
Arm/Group | Tramadol HCl OAD 200 mg | Tramadol IR (Ultram®) 50 mg 6-hourly
Number analyzed (Participants) | 26 | 26
percentage of fluctuation | 76.9 (20.0) | 91.1 (20.0)

6. Secondary Outcome: Percentage Swing
Description: Percentage swing is a pharmacokinetic parameter recommended by the FDA for submission and is calculated as follows:((Cmax,ss - Cmin,ss)/Cmin,ss)*100. It was calculated over 24 hours on day 5.
  Where:
  Cmax,ss = Maximum concentration at steady state; Cmin,ss = Minimum concentration at steady state.
Time Frame: 24 hours (day 5)
Measure: Mean (Standard Deviation); unit: percentage of fluctuation
Arm/Group | Tramadol HCl OAD 200 mg | Tramadol IR (Ultram®) 50 mg 6-hourly
Number analyzed (Participants) | 26 | 26
percentage of fluctuation | 131 (52) | 133 (40)

7. Secondary Outcome: Half-value Duration (HVD)
Description: Time over which plasma concentrations were above one half Cmax on day 5. 24h = 24 hours.
Time Frame: 24 hours (day 5)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tramadol HCl OAD 200 mg | Tramadol IR (Ultram®) 50 mg 6-hourly
Number analyzed (Participants) | 26 | 26
hours | 20.7 (2.56) | 22.0 (2.24)

8. Secondary Outcome: Plateau Time (T75%Cmax)
Description: Time over which plasma concentrations were above 75% Cmax on day 5. 24h = 24 hours.
Time Frame: 24 hours (day 5)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tramadol HCl OAD 200 mg | Tramadol IR (Ultram®) 50 mg 6-hourly
Number analyzed (Participants) | 26 | 26
hours | 11.5 (4.5) | 9.2 (3.3)

ADVERSE EVENTS:
Arm/Group | Tramadol HCl OAD 200 mg | Tramadol IR (Ultram®) 50 mg 6-hourly
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 12/26 | 10/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tramadol HCl OAD 200 mg (N=26) | Tramadol IR (Ultram®) 50 mg 6-hourly (N=26)
Constipation (Gastrointestinal disorders) | 4 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dry mouth (General disorders) | 2 (2) | 0 (0)
ALT elevated/raised (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Headache (General disorders) | 5 (5) | 3 (4)
Vomiting (Gastrointestinal disorders) | 3 (4) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a publication based on the results of this study is envisaged, approval from the sponsor will be obtained and a draft manuscript will be submitted to the sponsor for scrutiny and comment.